CLINICAL TRIAL: NCT03005977
Title: What Test is Most Sensitive in Identifying Stress Urinary Incontinence in Women With Pelvic Organ Prolapse; Urodynamics, Standing Cough Stress Test, or Pyridium Pad Test?
Brief Title: Identifying Stress Urinary Incontinence in Women With Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Eric Hurtado, Urogynecology Clinical Fellow, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FLA 16-078
Record Dates: First submitted 2016-12-15; First posted 2016-12-30 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Stress Urinary Incontinence; Pelvic Organ Prolapse
Keywords: Urodynamics; Pyridium pad test; Cough stress test; Pelvic organ prolapse
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Organ Prolapse | interventions — Urodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urodynamics, pyridium pad & cough stress (Other): The Pelvic Floor Bother Questionnaire, a questionnaire standardized by Cleveland Clinic Florida, the Urogenital Distress Inventory (UDI-6), and the numerical analog scale are to be administered prior to and 6 weeks after the surgical intervention. (14, 15)
  Prior to surgery, patients will be scheduled for a UDS performed by a qualified nurse practitioner or physician and will be given instructions in verbal and written form to undergo a 24 H pyridium pad test at least 72 hours before the UDS. Patients will be given pyridium TID and report if orange stain is noted on their pad in this period of time. A supine and a standing cough stress test will also be performed.
  Interventions: Procedure: Urodynamics

INTERVENTIONS:
Procedure: Urodynamics — UDS is to be performed with prolapse reduced by a speculum. The patient will be asked to valsalva three times then cough while seated after 150 ml of fluid is instilled in the bladder and then again at 300 ml. The same provocative measures will be performed at capacity, with the catheter in place and without the catheter if no leak is identified. If the patient leaks at any volume or if the patient leaks during the cough pressure profile (CPP), the test will be considered positive. If the patient does not leak during filling nor during the CPP then the test will be considered negative.
  Other Names: 24 hour pyridium pad test; Cough stress test

SUMMARY:
What test is most sensitive in identifying stress urinary incontinence in women with pelvic organ prolapse; urodynamics, cough stress test, or pyridium pad test? The hypothesis states that there is a difference between the sensitivity of UDS, pyridium pad test and cough stress tests, with UDS being the most sensitive and the gold standard in identifying SUI in patients with pelvic organ prolapse.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is the descent of the pelvic organs into or through the vagina. It is seen in about 11% of the female population by age 80 years old and is often treated with surgery. For patients with pelvic organ prolapse a complaint of de novo stress urinary incontinence (SUI), potential, or occult SUI after prolapse surgery is well-documented. This new onset of incontinence ranges from 6-60% of the time and therefore, patients who undergo surgery for POP are at risk for needing a subsequent procedure if SUI is not identified prior to the pelvic reconstruction.

Pre-operative evaluation for SUI includes a history and physical exam. The physical exam may include an empty supine stress test ESST, standing cough stress test (CST), pyridium pad test, and urodynamics (UDS). Prior studies have been performed to determine which of these tests are best at identifying SUI. One systemic review found that UDS was 92% sensitive in identifying SUI. When comparing UDS to the cough stress test and the weighed pyridium pad test, the cough stress test was found to be 90% sensitive and the pyridium pad test only 60% sensitive. The pyridium pad test was 68% sensitive when a pad test was found to be positive by orange color stain noted on the pad.

The various ways these tests are performed have also been evaluated. For example, there was no statistical difference in outcomes of a CST; whether completed supine or standing and independent of bladder volume. In regards to the pyridium pad tests, several studies have compared a 1 hour to 24 hour pyridium pad test with varying results of efficacy. Furthermore, in a study done when comparing pad weight and color, even asymptomatic women had positive pyridium pad tests suggesting this test is less specific in identifying SUI. A secondary analysis of the looked at how different reduction methods effect the predictability of post-operative SUI on UDS. Reduction of pelvic organ prolapse with a speculum was the most sensitive in identifying post-operative SUI at 53%. However, there is a paucity of evidence as to which pre-operative test is best in identifying SUI in patients with pelvic organ prolapse.

In this prospective study, the aim is to determine which test is most sensitive in pre-operatively identifying SUI and occult SUI in patients treated for prolapse. The hypothesis states that there is a difference between the sensitivity of UDS, pyridium pad test and cough stress tests, with UDS being the most sensitive and the gold standard in identifying SUI in patients with pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* 18 y/o or greater
* Able to consent
* Stage 2 or greater prolapse
* With or without complaint of stress urinary incontinence

Exclusion Criteria:

* Desire non-surgical management
* Prior surgery for prolapse or incontinence
* Treated medically for incontinence in the past 4 weeks
* Current Infection
* Known neurologic condition
* Stage 3 or greater chronic kidney disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with SUI as per Pelvic Floor Bother Questionnaire prior to prolapse surgery compared to number of patients with clinical SUI identified on either UDS, pyridium pad test and cough stress test. | 2 years
  Pelvic Floor Bother Questionnaire:A comparison will be made for each patient across the three studies to identify which test is most predictive of patient's SUI indicated by leakage identified on patients pre-operative questionnaire: Pelvic Floor Bother Questionnaire.
Number of patients with SUI as per the Urogenital Distress Inventory (UDI-6):Questionnaire prior to prolapse surgery compared to number of patients with clinical SUI identified on either UDS, pyridium pad test and cough stress test. | 2 years
  The Urogenital Distress Inventory (UDI-6):A comparison will be made for each patient across the three studies to identify which test is most predictive of patient's SUI indicated by leakage identified on patients pre-operative questionnaire: the Urogenital Distress Inventory (UDI-6)
Number of patients with SUI as per The numerical analog scale prior to prolapse surgery compared to number of patients with clinical SUI identified on either UDS, pyridium pad test and cough stress test. | 2 years
  The numerical analog scale.A comparison will be made for each patient across the three studies to identify which test is most predictive of patient's SUI indicated by leakage identified on patients pre-operative questionnaire: the numerical analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hurtado, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Data individual participant data will not be shared with other researches.

REFERENCES:
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] Latini JM, Kreder KJ Jr. Associated pelvic organ prolapse in women with stress urinary incontinence: when to operate? Curr Opin Urol. 2005 Nov;15(6):380-5. doi: 10.1097/01.mou.0000179760.45715.9b. PMID 16205487
- [Background] Kasturi S, Diaz SI, McDermott CD, Woodman PJ, Bump RC, Terry CL, Hale DS. De novo stress urinary incontinence after negative prolapse reduction stress testing for total vaginal mesh procedures: incidence and risk factors. Am J Obstet Gynecol. 2011 Nov;205(5):487.e1-4. doi: 10.1016/j.ajog.2011.07.006. Epub 2011 Jul 20. PMID 21925638
- [Background] Wei JT, Nygaard I, Richter HE, Nager CW, Barber MD, Kenton K, Amundsen CL, Schaffer J, Meikle SF, Spino C; Pelvic Floor Disorders Network. A midurethral sling to reduce incontinence after vaginal prolapse repair. N Engl J Med. 2012 Jun 21;366(25):2358-67. doi: 10.1056/NEJMoa1111967. PMID 22716974
- [Background] Brubaker L, Cundiff GW, Fine P, Nygaard I, Richter HE, Visco AG, Zyczynski H, Brown MB, Weber AM; Pelvic Floor Disorders Network. Abdominal sacrocolpopexy with Burch colposuspension to reduce urinary stress incontinence. N Engl J Med. 2006 Apr 13;354(15):1557-66. doi: 10.1056/NEJMoa054208. PMID 16611949
- [Background] Martin JL, Williams KS, Abrams KR, Turner DA, Sutton AJ, Chapple C, Assassa RP, Shaw C, Cheater F. Systematic review and evaluation of methods of assessing urinary incontinence. Health Technol Assess. 2006 Feb;10(6):1-132, iii-iv. doi: 10.3310/hta10060. PMID 16487456
- [Background] Price DM, Noblett K. Comparison of the cough stress test and 24-h pad test in the assessment of stress urinary incontinence. Int Urogynecol J. 2012 Apr;23(4):429-33. doi: 10.1007/s00192-011-1602-1. Epub 2011 Nov 16. PMID 22086265
- [Background] Reena C, Kekre AN, Kekre N. Occult stress incontinence in women with pelvic organ prolapse. Int J Gynaecol Obstet. 2007 Apr;97(1):31-4. doi: 10.1016/j.ijgo.2006.12.011. Epub 2007 Feb 8. PMID 17291508
- [Background] W. Henderson, S. Kane, J. Mangel, J. Garibay, E. Kikano, R. Pollard, S. T. Mahajan, A. Hijaz. A randomized comparative study correlating cough stress test with urodynamics and 24 hour pad test in the evaluation of stress urinary incontinence. J. Female Pelvic Medicine & Reconstructive Surgery Issue: September/October 2015. Volume 21(5) Supplement 1, p S11
- [Background] Artibani, W; Andersen, JT; Gajewski, JB; Ostergard, DR; Raz, S; Tubaro, A; Chapter 8C imaging and other Investigations. 2nd International Consultation on Incontinence 2002 p425-477
- [Background] Wall LL, Wang K, Robson I, Stanton SL. The Pyridium pad test for diagnosing urinary incontinence. A comparative study of asymptomatic and incontinent women. J Reprod Med. 1990 Jul;35(7):682-4. PMID 2198349
- [Background] Visco AG, Brubaker L, Nygaard I, Richter HE, Cundiff G, Fine P, Zyczynski H, Brown MB, Weber AM; Pelvic Floor Disorders Network. The role of preoperative urodynamic testing in stress-continent women undergoing sacrocolpopexy: the Colpopexy and Urinary Reduction Efforts (CARE) randomized surgical trial. Int Urogynecol J Pelvic Floor Dysfunct. 2008 May;19(5):607-14. doi: 10.1007/s00192-007-0498-2. Epub 2008 Jan 9. PMID 18185903
- [Background] Peterson TV, Karp DR, Aguilar VC, Davila GW. Validation of a global pelvic floor symptom bother questionnaire. Int Urogynecol J. 2010 Sep;21(9):1129-35. doi: 10.1007/s00192-010-1148-7. Epub 2010 May 11. PMID 20458467
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Derived] Martin L, Ossin D, Schachar J, Devakumar H, Alas A, Davila GW, Reis IM, Miao F, Hurtado E. Comparison of Methods to Identify Stress Urinary Incontinence in Women With Pelvic Organ Prolapse. Female Pelvic Med Reconstr Surg. 2021 Jan 1;27(1):e127-e132. doi: 10.1097/SPV.0000000000000858. PMID 33369965